CLINICAL TRIAL: NCT04523844
Title: Effect of Topical Prophylaxis With Brinzolamide-brimonidine Fixed Combination on Intraocular Pressure Elevation After Intravitreal Injections of Anti-vascular Endothelial Growth Factors
Brief Title: Brinzolamide-brimonidine Fixed Combination for Preventing IOP Elevation After Intravitreal Anti-VEGF Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Athens Elpis (Other)
Responsible Party: Principal Investigator, Maria Dettoraki, Locum Specialist, Department of Ophthalmology, General Hospital of Athens Elpis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1992
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Eye Diseases; Injection Complication; Intraocular Pressure
Keywords: anti-vascular endothelial growth factor; intraocular pressure; brinzolamide; brimonidine; fixed combination
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator who will measure the IOP will be masked to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brinzolamide-brimonidine fixed combination (Active Comparator): One drop of the brinzolamide-brimonidine fixed combination is instilled in the eyes of patients two hours before the intravitreal injection
  Interventions: Drug: Brinzolamide-brimonidine Fixed Combination
- No topical IOP-lowering medication (No Intervention): No IOP-lowering drops are instilled before the intravitreal injections

INTERVENTIONS:
Drug: Brinzolamide-brimonidine Fixed Combination — In case group one drop of a fixed combination of brinzolamide-brimonidine will be instilled two hours before the injection
  Other Names: Simbrinza 0.2%-1% Ophthalmic Suspension
  Arms: Brinzolamide-brimonidine fixed combination

SUMMARY:
This study aims to evaluate the effect of topical prophylaxis with brinzolamide-brimonidine fixed combination on short-term intraocular pressure (IOP) elevation after intravitreal injections of anti-vascular endothelial growth factors (anti-VEGF).

Patients scheduled for treatment with intravitreal injections of anti-VEGF will be randomly divided into two groups. In control group no prophylactic medication will be used, whereas in case group one drop of brinzolamide-brimonidine fixed combination will be instilled two hours before the injection. IOP will be measured before the injection, 1 minute after the injection, 10 minutes and 30 minutes post-injection in all eyes. In case group, the pre-injection IOP will be measured prior to the administration of the fixed combination of brinzolamide-brimonidine. The iCare (IC200) tonometer will be used for IOP measurements at all time points.

DETAILED DESCRIPTION:
The intravitreal anti-VEGF (ranibizumab, bevacizumab, pegaptanib and aflibercept) are commonly used in the treatment of diabetic macular edema, neovascular age-related macular degeneration and other pathologies characterized by retinal or choroidal neovascularization. Intravitreal injections οf anti-VEGF agents result in an immediate and transient increase in IOP, which returns to normal within a short period of time, typically within thirty minutes. Repeated intravitreal injections and prolonged treatments seem to be associated with sustained elevation of IOP, leading to the initiation of ocular hypotensive medication and glaucoma filtration surgery. A fixed-dose combination of brinzolamide 1%, a carbonic anhydrase inhibitor, and brimonidine 0,2%, an alpha 2 adrenergic receptor agonist, represents a safe and effective drug in glaucoma treatment and its ocular hypotensive effect has been demonstrated similar to or better than the unfixed combinations of its component drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for treatment with intravitreal injections of anti-vascular endothelial growth factors

Exclusion Criteria:

* history of glaucoma or ocular hypertension
* use of topical medications (e.g. IOP-lowering medication, corticosteroids)
* pseudoexfoliation
* pigment dispersion syndrome
* corneal diseases
* active intraocular inflammation
* any intraocular surgery in the last 6 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
IOP at 1 minute post-injection | 1 minute post-injection
  IOP will be measured by the same portable tonometer used before the injection (iCare-IC200 tonometer)

SECONDARY OUTCOMES:
IOP at 10 minutes post-injection | 10 minutes post-injection
  IOP will be measured by the same portable tonometer used before the injection (iCare-IC200 tonometer)
IOP at 30 minutes post-injection | 30 minutes post-injection
  IOP will be measured by the same portable tonometer used before the injection (iCare-IC200 tonometer)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dettoraki, MD, PhD, Principal Investigator — "Elpis" General Hospital of Athens
Locations (1):
- "Elpis" General Hospital, Athens, Ambelokipi, Greece